CLINICAL TRIAL: NCT07012564
Title: Does Vitamin C Improve Postoperative Healing: A Randomized Split-Mouth Clinical Trial After Impacted Mandibular Third Molar Surgery
Brief Title: Does Vitamin C Improve Postoperative Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Alper AKTAŞ, Professor, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HU-ADÇC-AA-01
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Impacted Mandibular Third Molar
Keywords: Vitamin C; Wound Healing; Third Molar Surgery; Oral Surgery; Postoperative Recovery; Trismus; Facial Swelling; Pain; Analgesic Use; Edema
MeSH Terms: conditions — Trismus; Pain; Edema | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This study employed a split-mouth crossover design, where each participant served as their own control. Bilateral surgical extractions of impacted mandibular third molars were performed in two separate sessions. The intervention (vitamin C) and the control (placebo) were randomly assigned to either the left or right surgical site, allowing intra-individual comparison of postoperative outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was designed as a double-blind trial. Both the participants and the outcome assessors were blinded to the allocation of the intervention (vitamin C or placebo). The tablets were identical in appearance, taste, and packaging to ensure blinding integrity. Allocation concealment was maintained by a third party responsible for randomization and distribution of the supplements. The clinical evaluator who performed the postoperative measurements (pain, swelling, trismus, and wound healing) was not informed about the intervention administered to each surgical site. Participants were also unaware of which side received vitamin C or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Patients received 1000 mg of oral vitamin C daily starting one day before surgery through postoperative day 7.
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Patients received an identical-looking placebo tablet once daily for the same duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000 mg oral vitamin C tablet taken daily from one day before surgery to postoperative day 7.
  Arms: Vitamin C
Other: Placebo — Identical-appearing oral tablet taken on the same schedule as the vitamin C group.
  Arms: Placebo

SUMMARY:
This randomized, split-mouth clinical trial investigates the effect of oral vitamin C supplementation on postoperative recovery following the surgical extraction of impacted mandibular third molars. Fifty-six healthy patients underwent bilateral extractions, with each side randomly assigned to receive either 1000 mg of oral vitamin C or a placebo. The supplementation began one day before surgery and continued through postoperative day 7. The outcome measures included facial swelling assessed through linear measurements (tragus-pogonion, tragus-commissure labiorum, and lateral canthus of the eye-angulus mandible), pain using a visual analog scale (VAS), trismus based on maximum interincisal opening, and early wound healing assessed with the Landry healing index. Analgesic consumption was also recorded. Pain was evaluated using VAS on days 1, 2, and 7. Edema, trismus, and early wound healing were evaluated on postoperative days 2 and 7. The study aims to determine whether vitamin C reduces edema, pain, and trismus, and enhances early soft tissue healing compared to placebo.

DETAILED DESCRIPTION:
This randomized, split-mouth clinical trial aimed to investigate the effect of oral vitamin C supplementation on postoperative recovery following the surgical extraction of impacted mandibular third molars. A total of 56 healthy patients requiring bilateral lower third molar extractions were included in the study. Each patient underwent two separate surgeries on both sides, with each side randomly assigned to receive either 1000 mg of oral vitamin C or a placebo.

Vitamin C supplementation started one day prior to surgery and continued for seven days postoperatively. The primary outcomes of the study were facial swelling, pain, trismus, and early soft tissue healing. Facial swelling was assessed using three linear measurements between specific anatomical landmarks: tragus-pogonion, tragus-labial commissure, and lateral canthus of the eye-angulus mandible. Trismus was measured based on maximum interincisal distance. Pain was evaluated using the visual analog scale (VAS) on postoperative days 1, 2, and 7. Edema, trismus, and early wound healing were assessed on postoperative days 2 and 7. Early wound healing was scored using the Landry healing index. Analgesic consumption was also recorded during the postoperative period.

This study was designed to evaluate whether vitamin C supplementation could reduce postoperative edema, pain, and trismus, and improve early soft tissue healing in comparison to placebo in the context of oral surgical procedures. The findings may provide evidence to support the use of vitamin C as an adjunctive therapy in oral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Systemically healthy
* Non-smoker
* No alcohol or substance abuse
* Bilateral impacted mandibular third molars
* Mesioangular impaction with a Pederson index of 5-6
* Voluntary participation
* Ability and willingness to attend follow-up visits

Exclusion Criteria:

* Pregnancy or lactation
* Presence of infection or pain related to third molars
* Associated pathological conditions (e.g., cysts or tumors)
* History of previous mandibular third molar extraction
* Congenital absence of third molars
* Known allergy to any drug or substance used in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Facial Swelling | Postoperative Day 2 and Day 7
  Facial swelling was measured using three linear distances: tragus-pogonion, tragus-labial commissure, and lateral canthus-mandibular angle.
Postoperative Pain Score (VAS) | Postoperative Days 1, 2, and 7
  Pain intensity was assessed using a 10-cm visual analog scale (VAS), with 0 = no pain and 10 = worst possible pain.

SECONDARY OUTCOMES:
Trismus (Maximum Interincisal Opening) | Postoperative Days 2 and 7
  Trismus was assessed by measuring the maximum interincisal distance in millimeters using a caliper.
Early Wound Healing (Landry Healing Index) | Postoperative Days 2 and 7
  Soft tissue healing was evaluated using the Landry healing index, which scores wound healing on a 5-point scale based on tissue color, bleeding, and granulation.
Analgesic Consumption | Postoperative Days 1,2 and 7
  : The number of analgesic tablets consumed was recorded for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No